CLINICAL TRIAL: NCT05883358
Title: Kratom Use Disorder Management Using Clonidine and/or Buprenorphine
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes2022 Kratom Addiction
Record Dates: First submitted 2023-05-03; First posted 2023-05-31 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Withdrawal Syndrome
Keywords: Kratom
MeSH Terms: conditions — Substance Withdrawal Syndrome | interventions — Clonidine; Buprenorphine

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kratom withdrawal: Kratom withdrawal syndrome patients, undergoing withdrawal therapy. On alternate weeks, each patient receives rotational treatment using Buprenorphine 5cmg/hr patch; or Clonidine tablet 0.1mg 4hourly; or combined Clonidine tablet 0.1mg 4hourly + Buprenorphine 5cmg/hr patch.
  Interventions: Drug: Clonidine, Buprenorphine

INTERVENTIONS:
Drug: Clonidine, Buprenorphine — Each patient receives rotational treatment using Buprenorphine 5cmg/hr patch; or Clonidine tablet 0.1mg 4hourly; or combined Clonidine tablet 0.1mg 4hourly + Buprenorphine 5cmg/hr patch.
  Other Names: Clonidine, Butrans

SUMMARY:
Kratom is used for stimulant, analgesic, anxiolytic, and sedative effects. There is inadequate knowledge about Kratom addiction. Kratom withdrawal may be treated like opioid withdrawal.

Prospective observational crossover study of consenting adults who are undergoing Kratom withdrawal management. On alternate weeks, each patient receives treatment using Buprenorphine 5cmg/hr patch; or Clonidine tablet 0.1mg 4hourly; or combined Clonidine tablet 0.1mg 4hourly + Buprenorphine 5cmg/hr patch. Each patient will undergo treatment for 12 weeks.

Patients will use Subjective Opiate Withdrawal Scale (SOWS) to collect data on daily basis. SOWS is a patient-administered tool that is used to record the severity and presence of opiate withdrawal. The physician will also use Clinical Opiate Withdrawal Scale (COWS) to collect data on weekly basis. COWS is a clinician-administered tool that is used to record the signs of opiate withdrawal. A change in the COWS and SOWS scores by 6-points is considered significant.

DETAILED DESCRIPTION:
Kratom herb is used for stimulant, analgesic, anxiolytic, and sedative effects. There is inadequate knowledge about Kratom dependence and withdrawal therapy. Kratom withdrawal may be treated with similar therapy for opioid withdrawal.

This is a prospective observational crossover study of consenting adult patients who are undergoing Kratom withdrawal management. On alternate weeks, each patient receives rotational treatment using Buprenorphine 5cmg/hr patch; or Clonidine tablet 0.1mg 4hourly; or combined Clonidine tablet 0.1mg 4hourly + Buprenorphine 5cmg/hr patch. Each patient will undergo Kratom withdrawal treatment for 12 continuous weeks.

The patient will use the Subjective Opiate Withdrawal Scale (SOWS), a special validated scale, to collect data on daily basis. The SOWS is a patient-administered tool that is used to record the severity and presence of opiate withdrawal symptoms. In addition, the physician will use the Clinical Opiate Withdrawal Scale (COWS), a special validated scale, to collect data on weekly basis. The COWS is a clinician-administered tool that is used to record the symptoms and signs of opiate withdrawal or substance abuse disorder. A change in the COWS and SOWS scores by 6-points is considered significant.

Data analyzed with IBM® SPSS® Statistics 25 (IBM Corp, Armonk, NY); using Student's t-test, ANOVA, Pearson Chi-square test, and regression analysis. P-value <0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

* adult patients
* Kratom dependence
* Kratom withdrawal syndrome
* Kratom withdrawal therapy
* good treatment compliance
* reliable Subjective Opiate Withdrawal Scale (SOWS) diary
* reliable Clinical Opiate Withdrawal Scale (COWS) diary
* informed consent for diary review
* consent for clinical record quality assurance review

Exclusion Criteria:

* poor treatment compliance
* cognitive disorder
* inability to provide consent
* major neuropsychiatric disorder
* unreliable diary
* cannabis use
* excessive alcohol intake
* previous adverse/allergic reactions to clonidine
* previous adverse/allergic reactions to buprenorphine

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients who have Kratom withdrawal syndrome; and undergoing medication treatment for Kratom withdrawal.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Opiate Withdrawal Score | 12 weeks
  Clinical Opiate Withdrawal Score on a scale of 5 to 36; low scores indicate mild withdrawal, high scores indicate severe withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Olu Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada